CLINICAL TRIAL: NCT05990998
Title: First Affiliated Hospital of Fujian Medical University
Brief Title: A Head-to-head Comparison of [68Ga]Ga-FAPI and [68Ga]Ga-TATE PET/CT in Patients With Nasopharyngeal Carcinoma: a Single-center, Prospective Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director of Nuclear Medicine Department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: First AHFujian
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Tumor Positron-Emission Tomography
MeSH Terms: interventions — gallium Ga 68 dotatate; 68Ga-FAPI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients will undergo a 68Ga-FAPI PET/CT and 68Ga-DOTATATE PET/CT (Experimental): NPC patients receive a single intravenous injection of 68Ga-FAPI PET/CT and 68Ga-DOTATATE PET/CT (2-4mCi) PET/CT,and undergo PET/CT scan at 40-60 min post-injection.
  Interventions: Drug: 68Ga-DOTATATE and 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-DOTATATE and 68Ga-FAPI — Each patient receive a single intravenous injection of 68Ga-FAPI or 68Ga-DOTATATE (2-4mCi) , and undergo PET/CT scan at 40-60 min post injection.

SUMMARY:
Both fibroblast activation protein (FAP)-targeted imaging and somatostatin receptors (SSTR)-targeted imaging were the promising imaging modalities for the diagnosis of primary and metastatic nasopharyngeal carcinoma (NPC). This prospective study is going to investigate to compare the diagnostic efficacy of 68Ga-FAPI and 68Ga-DOTATATE in detecting primary and metastatic NPC lesions, thereby obtaining a more accurate examination method of NPC.

DETAILED DESCRIPTION:
Patients with newly diagnosed or previously treated NPC will be recruited in this study.

Each patient received an intravenous injection of 68Ga-DOTATATE (2-4mCi) on the first day and 68Ga-FAPI (2-4mCi) on the second day. Whole-body PET/CT scans were performed at 40-60 min after injection on the same scanner. Physiologic normal-organ uptake, lesion numbers, and lesion uptake were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender, aged ≥ 18 years.

  * Patients with newly diagnosed or previously treated NPC
  * A diagnostic magnetic resonance imaging (MRI) of the tumor region within the previous 1 weeks prior to dosing day is available.
  * signed written consent.

Exclusion Criteria:

* pregnancy
* breastfeeding
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
SUVmax | through study completion, an average of 2 years
  Determination of SUV for detected lesions and discernible organs of 68Ga-FAPI and 68Ga-DOTATATE scan.
Lesion numbers | through study completion, an average of 2 years
  Determination of lesion numbers of 68Ga-FAPI and 68Ga-DOTATATE scan.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, M.D., Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No